CLINICAL TRIAL: NCT04160832
Title: Prevalence and Spectrum of Germline Cancer Susceptibility Gene Mutations Among Patients with Advanced Colorectal Polyps
Brief Title: Prevalence and Spectrum of Cancer Susceptibility Among Patients with Advanced Colorectal Polyps
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 18-2827.cc
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Neoplasm
Keywords: genetics; polyps; cancer; multi-gene panel
MeSH Terms: conditions — Colorectal Neoplasms; Polyps; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Genetic: Multi-Cancer Cancer Panel — Eligible patients will receive genetic testing to determine germline cancer predisposition.

SUMMARY:
The study is being conducted to determine the prevalence and risk factors for germline cancer susceptibility genetic mutations among patients with advanced colorectal polyps.

ELIGIBILITY:
Inclusion Criteria:

* Provision to sign and date the consent form
* Stated willingness to comply with all study procedures and be available for the duration of the study
* Be a male or female aged 18-89
* Undergone colonoscopy
* At least one advanced colorectal polyp, defined as having any of the following:
* Any polyp ≥ 1cm (adenoma or serrated polyp)
* Any polyp with villous architecture
* Any polyp with high-grade dysplasia
* Sessile serrated polyps with any dysplasia
* Traditional serrated adenoma

Exclusion Criteria:

* Known hereditary cancer syndrome
* Personal history of inflammatory bowel disease
* Personal history of colorectal cancer
* Polyp histology or size unavailable or not documented

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females aged 18 - 89, who have been diagnosed with advanced colorectal polyps.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of germline pathogenic/likely pathogenic variants in cancer predisposition genes in patients with advanced colorectal polyps | 3 years

SECONDARY OUTCOMES:
Risk factors for germline pathogenic/likely pathogenic variants in patients with advanced colorectal polyps | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Swati Patel, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No